CLINICAL TRIAL: NCT03992326
Title: Phase Ib Study To Assess The Feasibility And Safety Of Adoptive Transfer Of Autologous Tumor-Infiltrating Lymphocytes In Advanced Solid Tumors
Brief Title: Adoptive Transfer Of Autologous Tumor-Infiltrating Lymphocytes in Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Internal competitive study that is open
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, George Coukos, MD, PhD, Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-DO-0012-SolTIL_2018
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Cyclophosphamide; fludarabine; Interleukin-2; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TIL-ACT + LDI (Experimental): Non-myeloablative lymphodepleting chemotherapy (cyclophosphamide and fludarabine), Low Dose Irradiation (LDI), Tumor Infiltrating Lymphocyte (TIL)-Adoptive Cell Therapy (ACT), Interleukin-2 (IL-2).
  Interventions: Other: TIL; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2; Other: Radiotherapy

INTERVENTIONS:
Other: TIL — Adoptive transfer of Autologous Tumor-Infiltrating Lymphocytes
Drug: Cyclophosphamide — Cyclophosphamide will be administered as an intravenous (IV) infusion for two days.
Drug: Fludarabine — Fludarabine will be administered as an intravenous (IV) infusion for five days.
Drug: Interleukin-2 — After TIL infusion, IL-2 (optional) will be started as a bolus administration every eight hours, for a maximum of eight doses.
Other: Radiotherapy — Low-dose irradiation (1Gy) will be administered using tomotherapy to up to 20 measurable tumor lesions once before TIL infusion.

SUMMARY:
Single center, single arm phase Ib trial to test the feasibility and safety of Tumor- Infiltrating Lymphocyte-Adoptive Cell Therapy (TIL-ACT) combined with low-dose irradiation in patients with advanced or metastatic solid tumors. The trial is based on lymphodepleting chemotherapy followed by low dose irradiation (LDI), and then ACT utilizing ex vivo expanded TILs in combination with high dose IL-2 (optional, depending on patient's tolerance). LDI will be administered once to metastatic lesions using tomotherapy.

DETAILED DESCRIPTION:
The objective of the trial is to define the feasibility and safety of TIL-ACT in combination with low-dose irradiation (LDI) in patients with advanced or metastatic solid tumors.

Study treatment will begin with intravenous (IV) non-myeloablative (NMA) lymphodepleting chemotherapy composed by fludarabine and cyclophosphamide. Both treatments will be started on the same day. Fludarabine will be administered for five days, and cyclophosphamide for two days. Low-dose irradiation (LDI) will be then administered once, to up to 20 measurable tumor lesions using tomotherapy.

TIL infusion will be performed intravenously followed by high dose IL-2 administration every eight hours, for a maximum of eight doses. Supportive care will be given as needed during the whole treatment period.

Patients achieving a stable disease, partial response or complete response after TIL-ACT treatment will then enter a follow-up period for 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with locally advanced (not radically treatable) or metastatic solid tumors with the below cancer types, who progressed after at least one standard therapy for advanced disease, or for whom such therapy was proven to be intolerable, or is considered inappropriate. Prior immunotherapy is allowed.

   1. Breast cancer: irrespective of hormone receptor, Human epidermal growth factor receptor 2 (HER2) status or molecular subtype.
   2. Non-small cell lung cancer (NSCLC): irrespective of histological or molecular subtypes.
   3. Ovarian cancer: patients with high-grade serous ovarian cancer (HGSOC).
   4. Colon cancer: irrespective of molecular subtype.
   5. Other solid tumor: Patients with any other histology (any molecular subtype) with the exception of primary brain tumors, as well as cutaneous, mucosal, and ocular/uveal melanoma.
2. Patients who have previously undergone tumor resection or biopsy and for whom pre-REP TILs are already available and adequate for further REP expansion. The following conditions have to be met:

   a. The Manufacturing facility / sponsor representative confirms that adequate pre-REP material (in quantity and quality) is available to move to REP.
3. At least one lesion accessible to biopsy for translational research (TR) at baseline and D30, without putting the patient at unusual risk. Every effort should be made to obtain a fresh tumor biopsy upon enrolment, if previous collection of tissue is judged insufficient for study translational endpoints. The following exceptions are accepted for the baseline biopsy:

   a. Tumor material was properly collected for all protocol translational endpoints during harvesting surgery or biopsy for the TIL production (pre-REP) and no intercurrent anticancer therapy has been administered since that surgery or last biopsy. If patient has been treated with any antitumor therapy that may have altered the tumor microenvironment at the estimation of the PI, a repeat biopsy should be performed.
4. Male or female age ≥ 18 to ≤ 70 years at the time of informed consent. Patients aged >70 will be evaluated by the investigator, and decision will be made according to patient's status, upon agreement with the PI.
5. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) of 0 to 2.
6. Life expectancy of greater than 12 weeks.
7. Radiologically measurable disease (as per RECIST v1.1).

   1. Modified RECIST should be used for mesothelioma.
   2. Prostate Cancer Working Group 3 (PCWG3) criteria should be used for prostate cancer
8. Patients with brain metastases are eligible after discussion and agreement with the PI, provided there are no more than 3 residual metastases, that all metastases have been treated with stereotactic radiation therapy or gamma knife therapy and are asymptomatic. Lesions should be stable for at least 1 month, as determined by CT or MRI evaluation after treatment and should not require steroids.

   Note: Patients presenting between three and five treated and inactive brain metastases can be considered for enrollment, after discussion and agreement with the PI.
9. Adequate viral serology defined by the following laboratory results obtained during screening period (within 17 days prior registration).

   1. Seronegative for HIV infection (anti-HIV-1/-2)
   2. Seronegative for hepatitis B infection (HBsAg, total anti-hepatitis B core antigen (HBc), anti-HBs). Exception is made in case of prior vaccination. Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen HBsAg test and a positive anti-HBc antibody test) are eligible, if Hepatitis B virus (HBV) DNA test is negative.
   3. Seronegative for hepatitis C infection (anti-HCV): if a patient has positive anti-HCV antibody, a negative HCV RNA need to be obtained to register the patient.
10. Hematology

    1. Absolute neutrophil count ≥ 1.0 x 10^9 cell/L without the support of granulocyte colony stimulating factor (G-CSF).
    2. Platelet count ≥ 100 x10 ^9 cell/L
    3. Hemoglobin ≥ 80 g/L. Subjects may be transfused to reach this cut-off.
11. Coagulation

    a. International normalization ratio (INR) ≤1.5 times the upper limit of normal (x ULN) unless the subject is receiving anticoagulant therapy as long as INR/PT and partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants.

    i) Exception: for patients with hepatocellular carcinoma (HCC), the INR may be up to 2.2, as long as the Child-Pugh score is A6 maximum.

    b. PTT or activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless the subject is receiving anticoagulant therapy as long as INR/PT and PTT/aPTT is within therapeutic range of intended use of anticoagulants.
12. Chemistry:

    1. Serum Alanine transaminase (ALT)/Aspartate aminotransferase (AST) ≤ to 3 x ULN i) Exception: ALT/AST considered related to liver metastasis ≤ to 5 x ULN ii) Exception: for patients with HCC serum ALT/AST ≤ to 5 x ULN
    2. Total bilirubin ≤1.5 x ULN i) Exception: in patients with Gilbert's syndrome who must have a total bilirubin ≤2.5 x ULN ii) Exception: total bilirubin considered related to liver metastasis ≤3 x ULN iii) Exception: for patients with HCC total bilirubin ≤2.3 x ULN, as long as the Child-Pugh score is A6 maximum
    3. Creatinine clearance by Cockcroft-Gault formula ≥ 40 ml/min
13. Adequate cardiovascular function, with documented left ventricular ejection fraction (LVEF) ≥ 45%. This parameter must be documented within 12 weeks before registration
14. Adequate respiratory function with forced expiratory volume in 1 second (FEV1) ≥ 50% predicted, forced vital capacity (FVC) ≥ than 50% predicted and diffusing capacity of lung for carbon monoxide (DLCO) ≥ than 50% predicted corrected. Patients with lung cancer or mesothelioma and values slightly under these limits (but >30% of predicted) can be enrolled after discussion and approval by the trial chair. These parameters must be documented within 12 weeks before registration
15. At the time the patient receives the NMA chemotherapy regimen (D-7):

    1. ≥28 days must have elapsed from any chemotherapeutic cytotoxic drug
    2. ≥28 days must have elapsed from bevacizumab, aflibercept and other anti-angiogenic antibodies
    3. ≥28 days or 5 half-lives (whichever is shorter) must have elapsed from a non-cytotoxic drug including but not limited to trastuzumab, pertuzumab, and other molecular targeted therapy (such as tyrosine kinase inhibitors), etc… i) Note: In case of probable tumor flare upon stopping of the non-cytotoxic drug, the investigator may decide to shorten this delay, upon agreement of the trial chair, in a case-by-case approach.
    4. ≥21 days must have elapsed from the last antibody therapy that could affect an anti-cancer immune response, including but not limited to anti-CTLA4, anti-Programmed cell death protein 1 (PD-1)), anti-Programmed death-ligand 1 (PD-L1), anti-Tumor Necrosis Factor Receptor Superfamily, member 4 (OX-40), or anti-Lymphocyte-activation gene 3 (LAG3) antibody therapy or their combination
    5. Exceptions: denosumab and biphosphonates are permitted
    6. Exceptions: androgen-deprivation therapy (ADT) for prostate cancer and hormonal therapy for breast cancer are permitted (and will be administered as SOC).
16. Patients' toxicities from previous therapies must have recovered to at least grade 1 according to NCI CTCAE v5.0, except for toxicities described below, as long as they do not put at risk the patient's condition and do not require systemic immunosuppressive steroids at immunosuppressive doses, including but not limited to:

    * Fatigue
    * Alopecia
    * Skin disorders
    * Stable neuropathy
    * Endocrinopathies requiring replacement treatment Note: For other medical conditions, or for any other toxicity with a higher grade but controlled by adequate treatment, prior discussion and agreement with the trial chair is mandatory.

    Note: Patients may have undergone surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less.
17. For women of childbearing potential (WOCBP: sexually mature women who have not undergone a hysterectomy and/or bilateral oophorectomy, have not been naturally post-menopausal for at least 12 consecutive months or have a serum follicle-stimulating hormone (FSH) < 40 milli-international units per milliliter (mIU/ml):

    1. Agreement to follow instructions for method(s) of contraception for the couple from screening until month 6 post start of NMA chemotherapy of the study.
    2. Negative pregnancy test (urine or serum) during screening.
18. For men participating in the trial and their female partners: agreement to follow instructions for method(s) of contraception for the couple from screening until month 6 post start of NMA chemotherapy of the study.

Exclusion Criteria:

1. Patients with an active second malignancy, except for

   1. non-melanoma skin cancer that has been apparently cured or successfully resected
   2. carcinoma in situ as long as they have been adequately treated
   3. Any malignancy that can be adequately managed expectantly without compromising prognosis, and after PI agreement..

   Patients who have a history of malignancy are not considered to have an active malignancy if they have completed therapy since at least 2 years and are considered by their treating investigator to be at ≤ 30% risk for relapse.
2. Patients with known peritoneal metastases who have a recent history of intermittent bowel obstruction (even partial), unless such obstruction has been resolved. Agreement with the Trial Chair is mandatory.
3. Patients with leptomeningeal carcinomatosis
4. History of idiopathic pulmonary fibrosis or evidence of active pneumonitis (any origin)
5. History of recent myocardial infarction or unstable angina, either within six months of enrolment
6. Documented Child-Pugh score of B or C for hepatocellular carcinoma patients with known underlying liver dysfunction
7. Active severe systemic infections within four weeks prior to beginning of NMA chemotherapy.
8. Patient requiring regular systemic immunosuppressive therapy (for example for organ transplantation, chronic rheumatologic disease); all immunosuppressive medications including but not limited to steroids, mycophenolate mofetil, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (TNF)-alpha agents must have been discontinued within the last two weeks prior to starting NMA chemotherapy.

   1. Note: Use of inhaled or topical steroids or corticosteroid use for radiographic procedures is permitted
   2. Note: The use of physiologic corticosteroid replacement therapy is permitted.
9. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
10. History of immediate hypersensitivity reaction to aminoglycosides (e.g. gentamicin or streptomycin).
11. Women who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
12. Subjects for whom there are concerns that they will not reliably comply with the requirements for contraception should not be enrolled into the study.
13. Any serious underlying medical condition that could interfere with study medication and potential adverse events.
14. Any mental or other impairment that may compromise compliance with the requirements of the study.
15. Patient participation in any other study currently receiving treatment. If the patient is in the follow-up period, he/she may be enrolled, as far as the elapsed time since the last previous treatment administration and the preparative regimen (NMA chemotherapy) is respected according to Inclusion Criteria n°15).
16. Participation in a research project using radiation sources exceeding an effective dose of 5 millisievert (mSv) with no direct benefit within the 12 last months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of TIL-ACT in combination with LDI - successful Rapid Expansion Protocol (REP): Number of patients for whom TIL cultures | Evaluated for each patient at day 0. After day 0 of the last patient, the number of patients with successful TIL-ACT infusion will be calculated.
  Number of patients for whom TIL cultures after REP achieve the required cell number and release criteria to start TIL-ACT infusion.
Feasibility of TIL-ACT in combination with LDI - successful infusion: Number of patients receiving a complete TIL-ACT infusion | Evaluated for each patient at day 0, up to 60 mins after start of TIL-ACT infusion. At day 0 of the last patient, the number of patients with successful TIL-ACT infusion will be calculated.
  Number of patients receiving a complete TIL-ACT infusion (planned NMA chemotherapy, planned LDI and at least partial TIL infusion; no minimum IL-2 required)
Toxicity of TIL-ACT and LDI | Treatment limiting toxicity (TLT) period: from chemotherapy start until Day30
  Number of patients with adverse events as assessed by CTCAE version 5.0

SECONDARY OUTCOMES:
Disease control rate (DCR) | 1, 3, 6, 9, 12 months
  Achievement of complete response, partial response or stable disease
Objective response rate (ORR) | 1, 3, 6, 9, 12 months
  Best overall response
Progression free survival (PFS) for TIL-ACT | 5 years
  Time from start of NMA chemotherapy until objective tumor progression (using RECIST criteria) or death if not documented progression.
Overall survival (OS) | 5 years
  Time from start of NMA chemotherapy until death

CONTACTS AND LOCATIONS:
Overall Officials: George Coukos, MD, PhD, Principal Investigator — Department director
Locations (1):
- CHUV Oncology Department, Lausanne, Canton of Vaud, Switzerland